CLINICAL TRIAL: NCT04512430
Title: A Phase II Trial of Neoadjuvant Treatment Carboplatin-Pemetrexed-Bevacizumab Plus Atezolizumab for the Treatment of Locally Advanced and Potentially Resectable NSCLC Patients With EGFR Mutations
Brief Title: Neo-DIANA: Neoadjuvant Treatment for EGFR Mutated Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP 20/01_Neo-DIANA; 2020-000642-33 (EudraCT Number)
Record Dates: First submitted 2020-08-07; First posted 2020-08-13 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Non Small Cell Lung Cancer; EGFR Gene Mutation
Keywords: Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Lung Diseases; Carcinoma, Bronchogenic; Carcinoma, Non-Small-Cell Lung; Bronchial Neoplasms; Atezolizumab; Bevacizumab; Carboplatin; Pemetrexed; Neoadjuvant treatment; Adjuvant treatment; Antineoplastic Agents, Immunological; EGFR Mutation; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Lung Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms | interventions — atezolizumab; Bevacizumab; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Neo-Adjuvant Immunotherapy (Experimental): * Neoadjuvant treatment: (Atezolizumab: 1200 mg, IV infusion+Bevacizumab: 15mg/Kg mg, IV infusion+Carboplatin: AUC6, IV infusion+Pemetrexed: 500 mg/m2, IV infusion) will start within 1-3 days from enrollment. 3 cycles will be administered at 21-day (+/- 3 days) intervals (QW3) prior to surgery.Before surgery a tumor assessment will be done. Patients must leave the study if there is evidence of progression. Patients with stable disease or partial response may be considered for surgery.
  * Surgery: Surgery must be done within the 4th week (+7 days) from day 21 cycle 3 of neoadjuvant treatment (day 42-49 after day 1 of cycle 3).
  * Adjuvant treatment: Atezolizumab: 1200 mg, IV infusion Q4W (+/- 3 days) for 6 months (6 cycles) Patients that are R0 confirmed by surgical pathology evaluation will receive the first adjuvant administration within the 3rd to 8th week (+7 days) from surgery and for 6 months (6 cycles).
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Atezolizumab — Patients will receive 1200 mg of Atezolizumab every 21 days (QW3) (+/- 3 days) during neoadjuvant phase and every 28 days (QW4) (+/- 3 days) at adjuvant phase in a monitored setting where there is immediate access to trained personnel and adequate equipment/medicine to manage potentially serious reactions.
  First Infusion
  * No premedication administered for atezolizumab specifically is permitted
  * Infuse atezolizumab (1200 mg in a 250 mL 0.9% NaCl IV bag) over 60 (+/- 15) minutes.
  Subsequent Infusions:
  * If patient experienced infusion-related reaction during any previous infusion, premedication with antihistamines may be administered for Cycles > 2 at the discretion of the treating physician.
  * If the patient tolerated the first infusion well without infusion-associated adverse events, the successive infusion may be delivered over 30 (+/- 10) minutes.
  Other Names: Tecentriq
Drug: Bevacizumab — Patients will receive 15mg/Kg of Avastin® (bevacizumab) administered by IV infusion every 21 days, for 3 cycles during neoadjuvant phase, in a monitored setting where there is immediate access to trained personnel and adequate equipment/medicine to manage potentially serious reactions.
  Other Names: Avastin
Drug: Carboplatin — Structure: The cis-diamino (cyclobutan-1, 1 dicarboxilate) platin. Stability: 24 hours at ambient temperature in 5% glucose, glucosaline or physiologic saline. It is recommended not to dilute with chlorinated solutions since this could affect the carboplatin.
  Route of administration: Intravenous infusion Patients will receive Carboplatin AUC6 administered by IV infusion every 21 days, for 3 cycles during neoadjuvant phase.
  Guidelines of Carboplatin administration: According to the standard of each center
  Other Names: Paraplatin
Drug: Pemetrexed — Patients will receive Pemetrexed 500mg/m2 administered by IV infusion every 21 days, for 3 cycles during neoadjuvant phase.
  Pemetrexed disodium (ALIMTA®, pemetrexed) is a novel pyrrolo[2,3 d]pyrimidine-based folic acid analogue.
  Route of administration: Intravenous infusion. Guidelines of Pemetrexed administration: According to the standard of each center
  Other Names: Alimta

SUMMARY:
This is an open-label, non-randomised, phase II, multi-centre clinical trial

26 patients will be enrolled in this trial to evaluate the major pathologic response in patients with neoadjuvant treatment with Carboplatin Pemetrexed Bevacizumab plus Atezolizumab in patients with non-small cell lung carcinoma locally advanced mutated in EGFR

DETAILED DESCRIPTION:
This is an open-label, non-randomised, phase II, multi-centre clinical trial. Patients enrolled will receive Atezolizumab 1200mg + Bevacizumab 15mg/Kg + Carboplatin AUC6 + Pemetrexed 500mg/m2 for 3 cycles every 21 days (+/- 3 days) as neoadjuvant treatment followed by surgery and 6 months of adjuvant treatment with Atezolizumab 1200 mg Q4W (+/- 3 days).

The primary objective is to evaluate the major pathologic response defined as 10 percent or fewer viable cancer cells detectable in the resected tumor and in lymph nodes in stage IIIA EGFR mutated patients treated in neoadjuvant setting with atezolizumab- bevacizumab- carboplatin and pemetrexed.

Patient accrual is expected to be completed within 2 years excluding a run-in-period of 3-6 months. Treatment and follow-up are expected to extend the study duration to a total of 6 years. Patients will be followed 3 years after adjuvant treatment. The study will end once survival follow-up has concluded. This will be followed by a close out period of 4 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. Previously untreated patients with histologically- or cytologically- documented NSCLC who present stage IIIA disease (according to 8th version of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology). PET/CT including IV contrast (CT of diagnostic quality) will be performed at baseline (28 days +10 before randomization).
* 2. Tumor should be considered resectable before study entry by a multidisciplinary team
* 3. Sensitizing EGFR mutation (Del Exon 19 and ins Exon 21).
* 4. ECOG (Performance status) 0-1
* 5. Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to randomization i. Neutrophils ≥ 1500×109/L ii. Platelets ≥ 100 ×109/L iii. Hemoglobin > 9.0 g/dL iv. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below): a. Female CrCl = (140 - age in years) x weight in kg x 0.85/ 72 x serum creatinine in mg/dL b. Male CrCl = (140 - age in years) x weight in kg x 1.00/ 72 x serum creatinine in mg/dL v. AST/ALT ≤ 3 x ULN vi. Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL) vii. PT/APTT/INR within normal limits
* 6. Measurable or evaluable disease according to RECIST v1.1.
* 7. The patients need to have a forced expiratory volume (FEV1)≥ 1.2 liters or >40% p- predicted value.
* 8. All patients are notified of the investigational nature of this study and signed a written informed consent in accordance with institutional and national guidelines, including the Declaration of Helsinki prior to any trial-related intervention.
* 9. Patients aged > 18 years.
* 10. Patient capable of proper therapeutic compliance and accessible for correct follow-up.
* 11. For female patients of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate (< 1% per year) when used consistently and correctly, and to continue its use for 5 months after the last dose of Atezolizumab and/or 6 months after the last dose of Bevacizumab, whichever is later. Such methods include: combined (estrogen and progestogen containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation together with another additional barrier method always containing a spermicide, intrauterine device (IUD): intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner (on the understanding that this is the only one partner during the whole study duration), and sexual abstinence.
* 12. For male patients with female partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate [< 1% per year] when used consistently and correctly, and to continue its use for 6 months after the last dose of Bevacizumab. Male patients should not donate sperm during this study and for at least 6 months after the last dose of Bevacizumab.
* 13. Oral contraception should always be combined with an additional contraceptive method because of a potential interaction with the study drugs. The same rules are valid for male patients involved in this clinical study if they have a partner of childbirth potential. Male patients must always use a condom.
* 14. Women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 14 days prior to initiation of study drug

Exclusion Criteria:

* 1. All patients carrying other EGFR mutations.
* 2. Patients with known anaplastic lymphoma kinase (ALK) fusion oncogene, STK11 ligand alteration or ROS1 translocations.
* 3. Clinically significant comorbidities that impaired administration of platinum-based chemotherapy.
* 4. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* 5. Patients with a history of interstitial lung disease cannot be included if they have symptomatic ILD (Grade 3-4) and/or poor lung function. In case of doubt please contact trial team.
* 6. Patients with other active malignancy requiring concurrent intervention and/or concurrent treatment with other investigational drugs or anti-cancer therapy.
* 7. Patients with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period.
* 8. Any medical, mental or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or understand the patient information.
* 9. Patients with positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
* 10. Patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* 11. Active tuberculosis.
* 12. Severe infections within 4 weeks prior to be included in the study, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
* 13. Patients with history of allergy to study drug components excipients.
* 14. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* 15. Women who are pregnant or in the period of breastfeeding.
* 16. Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the study.
* 17.

  * Patients with active, known or suspected autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
  * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for this study.
  * Patients with controlled Type 1 diabetes mellitus on a stable dose of insulin regimen are eligible for this study.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * Rash must cover less than 10% of body surface area (BSA).
    * Disease is well controlled at baseline and only requiring low-potency topical steroids.
    * No acute exacerbations of underlying condition within the previous 12 months (not requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high-potency or oral steroids).
* 18. Patients with any contraindication for bevacizumab administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Principal Investigator — Hospital Puerta del Hierro
Locations (18):
- Spain (18):
  - ICO Badalona, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - ICO Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Insular de Gran canaria, Las Palmas de Gran Canaria, Gran Canaria
  - Complejo Hospitalario de Navarra, Pamplona, Iruña
  - Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Universitari Quiron Dexeus, Barcelona
  - Hospital Universitari Vall d' Hebron, Barcelona
  - ICO Girona, Hospital Josep Trueta, Girona
  - Hospital Universitario de Jaén, Jaén
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital General Universitario de Málaga, Málaga
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Neo-Adjuvant Immunotherapy: Neoadjuvant treatment: (Atezolizumab: 1200 mg, IV infusion+ Bevacizumab: 15mg/Kg mg, IV infusion+Carboplatin: AUC6, IV infusion+ Pemetrexed: 500 mg/m2, IV infusion) will start within 1-3 days from enrollment. 3 cycles will be administered at 21-day intervals (QW3) prior to surgery.Before surgery a tumor assessment will be done. Patients must leave the study if there is evidence of progression. Patients with stable disease or partial response may be considered for surgery.
  Surgery: Surgery must be done within the 4th week
  Adjuvant treatment: Atezolizumab: 1200 mg, IV infusion Q4W for 6 months (6 cycles) Patients that are R0 confirmed by surgical pathology evaluation will receive the first adjuvant administration within the 3rd to 8th week from surgery and for 6 months (6 cycles).
Period: Overall Study
Arm/Group | Experimental: Neo-Adjuvant Immunotherapy
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: Neo-Adjuvant Immunotherapy
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 66.5 [51 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Spain | 4
Smoking status [Count of Participants; unit: Participants]
  Never smoker (<= 100 cigarettes/lifetime) | 3
  Former smoker (>= 1 year) | 1
  Active smoker | 0
Performance status [Count of Participants; unit: Participants] — ECOG Performance Status Scale: It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability
  GRADES:
  ECOG 0: Fully active. ECOG 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours ECOG 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours ECOG 4: Completely disabled ECOG 5: Dead
  Participants
    ECOG 0 | 2
    ECOG 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: To determine the antitumor activity in terms of objective response rate (ORR) of neoadjuvant treatment with carboplatin-pemetrexed-bevacizumab plus atezolizumab for the treatment of locally advanced and potentially resectable NSCLC patients with EGFR mutations.
  Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Progressive disease (PD): at least a 20% increase in the sum of diameters of target lesions.
Time Frame: From date of end of neoadjuvant treatment until the date of last follow up, assessed up to 36 months
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Neo-Adjuvant Immunotherapy
Number analyzed (Participants) | 4
Participants
  Partial Response (PD) | 1
  Stable Disease (SD) | 2
  Progression Disease (PD) | 1

ADVERSE EVENTS:
Time Frame: 40 months
Arm/Group | Experimental: Neo-Adjuvant Immunotherapy
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Neo-Adjuvant Immunotherapy (N=4)
Right lung hernia (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Neo-Adjuvant Immunotherapy (N=4)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
COVID 19 (Infections and infestations) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The recruitment was closed prematurely to due to slow recruitment, so there are no consistent data to achieve any relevant conclusion at this point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT04512430/Prot_SAP_000.pdf